CLINICAL TRIAL: NCT04151862
Title: Therapeutic Contact Lenses vs. Tight Bandage Patching and Pain Following Pterygium Excision: a Prospective Randomized Controlled Study
Brief Title: The Two Most Common Ways Post-operative Eye Patch Are Therapeutic Contact Lenses (TCL) and Overnight Bandaging With Tight Bandage Patch: This Study is Designed to Determine the Most Effective Post-operative Care to Relief the Patient's Discomfort After Pterygium Excision Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Dr Erez Tsumi, Head of Ophthalmology Department, Soroka University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0145-19 SOR
Record Dates: First submitted 2019-10-27; First posted 2019-11-05 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Pterygium of Both Eyes; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tight eye bandage (Active Comparator): Both eyes will be operated at two separate sessions. In the first session the first 25 patients will be bandaged postoperatively with tight eye bandage patching.
  Interventions: Device: tight eye bandage
- therapeutic contact lenses (TCL) (Active Comparator): Both eyes will be operated at two separate sessions. In the second session the 25 patients will be bandaged postoperatively with therapeutic contact lenses (TCL).
  Interventions: Device: Soflex Soft Contact Lens

INTERVENTIONS:
Device: tight eye bandage — sterile eye pad made of 100% cotton
  Other Names: Nissan LTD
  Arms: tight eye bandage
Device: Soflex Soft Contact Lens — Therapeutic contact lenses (TCL)
  Other Names: SOFLEX LTD (TH78)
  Arms: therapeutic contact lenses (TCL)

SUMMARY:
This study is designed to determine the most effective post-operative care to relief the patient's discomfort after pterygium excision surgery.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled trial. 50 patients with primary pterygium in both eyes for whom surgery was advised, will be recruited to the study. Criteria for pterygium excision surgery is mostly cosmetic, local eye symptoms, or visual impairment.

The following data will be collected and analyzed:

1. Demographic data such as: age, gender
2. Clinical data: best-corrected visual acuity (BCVA) full biomacroscopy examination, before surgery and at post-operative day (POD) 1 and 3
3. Symptoms and discomfort: Visual Analogue Scale (VAS) score and pain killer use. The differences in these variables values preoperatively and on the first and 3rd postoperative day will compared between the two treated eyes.

Surgical technique and postoperative care

All patients will be operated for the same pterygium excision under local anesthesia in the formal accepted surgical method. All patients will be treated with ofloxacin drops + dexamethasone drops four times daily during the first postoperative week. The only difference is that one group will be bandaged with tight bandage patching and the other with therapeutic contact lenses (TCL) only for the first 24 hours.

Patient-centered outcome

Discomfort and pain will be evaluated on the follow-up meeting on the first and 3rd postoperative day. The patient will be asked to rate pain and discomfort for each operated eye on pain scale of VAS ranking the pain on a line from No pain at 0 cm to worst possible pain at 10 cm and the estimated pain given by the patient's translation of pain into spot on a line.

Patients will also be queried about the number of hours during which they feel pain, and the number of pain killers used ( every patient will be given prescription for 3 tabs of Paracetamol 500 mg (giving no drugs sensitivity for paracetamol) on POD 1 & 3).

Their sleep quality will rated according to whether they reported having a full night's sleep and the number of times they were awoken due to pain/discomfort.

Statistical analysis

The t test was used to calculate differences in numerical variables (VA, hours of pain, number of pain killers, etc.). Non-parametric Wilcoxon Mann-Whitney was used to calculate differences in non-numerical variables such as pain level (VAS scale). Chi-square analyses were used to calculate proportional group differences (e.g., use of pain killers and sleep pattern). The overall significance level was set to a value of 0.05. The statistical analysis was carried out using Microsoft Excel 2013.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients with no significant ocular diseases, older than 18 year old with both eyes pterygia, referred for surgery and which are interested of their own will for pterygium excision surgery.

Exclusion Criteria:

* patients younger than 18 years old
* patients with chronic diseases of the immune system
* chronic diseases of eyelid or ocular surface, history of previous ocular surgery or trauma
* collagen vascular disease or diabetes mellitus chronic
* ingestion of pain killers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Measurment of pain and discomfort for patients post pterygium excision: Visual Analog Scale by questionnaire on marking straight horizontal line of fixed length from 0-100 mm where 0 mm is no pain and 100 mm is maximal pain. | 1st Post Operative Day and 3rd Post Operative Day
  Assessing pain and discomfort comparing the two groups ( one with tight bandage and the other with contact lens).post pterygium excision by the change in pain scores on Visual Analog Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Erez Tzumi, MD, Principal Investigator — Head of ophthalmology department

IPD SHARING:
Plan to Share IPD: No